CLINICAL TRIAL: NCT04743648
Title: Effect of The Innovatıve Thınkıng Development Program on The Innovatıve Approaches, Crıtıcal Thınkıng and Perceıved Competence of Nursıng Students
Brief Title: Effect of Innovative Thinking Development Program on Some Approaches of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ilknur Aydin Avci, Professor, Ondokuz Mayıs University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019/340
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Program Development; Educational Problems
Keywords: creativity; critical thinking; innovative thinking; nursing education; nursing students

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group (Experimental): After determining the experimental and control groups, pre-tests were performed.The program was applied to students in the experimental group.The program was implemented for six weeks based on the theme of innovative thinking.The program developed a training program based on the Tyler Taba model. This model, which is often used in developing educational programs, includes all the necessary steps to teach and accept a new concept. In the ITDP training program, an interactive educational content has been created in which knowledge will be transformed into behavior.In the training, subjects were taught in units, workshops were held, seminars were given. Post-tests were applied at the end of the training.
  Interventions: Behavioral: Innovative Thinking Development Program (ITDP)
- Control Group I (No Intervention): Pre-test and post-tests were applied to the non-intervention group
- Control Group II (No Intervention): Pre-test and post-tests were applied to the non-intervention group

INTERVENTIONS:
Behavioral: Innovative Thinking Development Program (ITDP) — With the implementation of the program, nursing students are expected to develop innovative thinking skills.
  Arms: Intervention Group

SUMMARY:
Background: This study was conducted to determine the effect of the Innovative Thinking Development Program (ITDP) on the innovative approaches, critical thinking and perceived competence of nursing students.The study has a non-randomized, control group pre-test-post-test experimental research design. The study population consisted of senior students in the Nursing Department of two similar faculties in the academic calendar 2019-2020 (n=164). In the study, the ITDB developed by the researcher was applied to the students in the experimental group. The research data were collected online using a 'Personal Information Form', 'Individual Innovativeness Scale', 'Marmara Critical Thinking Trends Scale', 'Self-Efficacy Scale' and 'Success Test 'developed by the researcher. Independent samples t test, Kruskal Wallis, Wilcoxon, ANOVA tests were used in the analysis of the data. Institutional permissions and ethics committee approval was obtained for the research.

Hypothesis:

H0: The innovative approaches, critical thinking tendencies and competence perceptions of nursing students included in ITDP do not change.

H1: Individual innovativeness, critical thinking disposition and self-efficacy scale scores of nursing students in the experimental group will change after ITDP.

DETAILED DESCRIPTION:
This study was conducted to determine the effect of the ITDP on the innovative approaches, critical thinking and perceived competence of nursing students.The non randomized clinical trial was based on the guidelines proposed by the Consolidated standard of Reporting Trials- CONSORT 2010. The data of the research were collected in Giresun and Ordu University Health Science Faculty between April 2020- October 2020.

In this study, there is a non-randomized experimental group and two control groups (total 164 nursing students). Experimental and control groups were determined by lots. Data collected through online forms.

The developed educational program was implemented to students in the experimental group through an online platform. The trainings lasted 6 weeks and different applications were made with themes appropriate to the content. In addition, a whatsapp group was opened and posts about innovation thinking exercises were made.

The research data were collected a 'Personal Information Form', 'Individual Innovativeness Scale', 'Marmara Critical Thinking Trends Scale' and 'Self-Efficacy Scale' in pre test and post tests.The efficiency of the program was determined by applying an 'Success Test' to the experimental group.

Personal Information Form: The twenty-one question 'Personal Information Form' consists of sociodemographic questions and questions related to innovation.

Individual Innovation Scale (IIS): The scale was developed in 1977. The scale was adapted to Turkish in 2014. The scale adapted to nursing is 5-point Likert type. It consists of three sub-dimensions and a total of 18 questions. These sub dimensions are; resistance to change sub-dimension, opinion leadership sub-dimension and risk-taking sub-dimension. According to the score obtained from the scale; Scores of 57 and below are classified as 'traditionalist', those who score between 58-65 as 'skeptical', those who score between 66 and 74 as 'questioning', those who score between 75 and 82 as 'pioneer', and those who score 82 and above as 'innovative'. Scale Cronbach Alpha value is 0.82. The Cronbach Alpha value of the scale for this study is 0.94.

Marmara Critical Thinking Trends Scale (MCTTS): The scale was developed in 2018. The scale consists of 28 items and 6 sub-dimensions. The scale is in 5-point Likert type. Scale sub-dimensions; reasoning, reaching judgment, searching for evidence, searching for truth, open-mindedness and systematicity. The high score obtained from each sub-dimension of the scale indicates that the individual has the feature in the relevant sub-dimension. Scale Cronbach Alpha value is 0.91. The Cronbach Alpha value of the scale for this study is 0.93.

Self-Efficacy Scale (SES):The scale was developed in 1983.The scale was adapted to Turkish in 1999. It is a 5-point Likert type consisting of 23 items. The 4 sub-dimensions of the scale are starting behavior, maintaining behavior, completing behavior and struggling with obstacles. The high total score obtained from the scale indicates that the general efficacy perception is high, and the low general efficacy perception is low. Scale Cronbach Alpha value is 0.81. The Cronbach Alpha value of the scale for this study is 0.88.

Evaluation of Data SPSS 23.0 statistical package program was used for statistical analysis and evaluation of the data. Whether the data showed normal distribution was checked with the Kolmogorov-Smirnov test. Independent samples t test and Mann Whitney U test were used to compare data between groups according to normality test. Paired samples t test and Wilcoxon test were used to compare the pre-test and post-test values within the group. The Chi-square test and two ratio tests were used to analyze categorical data. Significance level was taken as p <0.05.

Information:

No budget was received from any institution for the research. Ethics committee approval was obtained and verbal consent was obtained from the participants.

There is no conflict of interest.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being open to communication,
* Being a fourth year nursing student,
* Not to be an innovation and entrepreneurship course in the curriculum,
* Students have online access opportunities.

Exclusion Criteria:

* Not being willing to participate in the study,
* Not being open to communication,
* Not being a fourth year nursing student,
* To come by undergraduate transfer and to have taken innovation and entrepreneurship course at the faculty he came from,
* Students do not have online access facilities.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Individual Innovativeness Scale | 3 months
  The scale measures individual innovativeness level. The lowest 18 points on the scale and 90 points are the highest. Based on the score obtained from the scale; 57 points and six fields 'traditionalist', 58-65 points to the areas between the 'skeptic', 66-74 score between 'questioner', 75-82 score between 'pioneer', those who scored above 82 points and 'innovative' are classified as.The increase in the scores obtained from the scale shows that the people are innovative.
Critical Thinking Trends Scale | 3 months
  The scale measures people's tendency to think critically. A high score taken from each sub-dimension indicates that the individual has a characteristic of the corresponding sub-dimension, and a total critical thinking trends score is obtained from the scale. The higher the score, the higher the critical thinking disposition.The highest score on the scale is 140.
Self-Efficacy Scale | 3 months
  This scale is used to measure people's perceptions of competence. Scores between 23 and 115 can be obtained from the scale. A high overall score on the scale indicates that people's overall perception of competence is high, and a low overall perception of competence is low.
Success Test | 3 months
  The test, developed in accordance with innovative thinking skills, consists of 20 questions.The highest 20 points and the lowest 0 points are taken from this test. The higher the score, the higher the innovative thinking.This test was developed to test the effectiveness of the training program on innovative thinking and to evaluate students' success on this subject. Pre-test was applied to the experimental group as post-test.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur Aydın Avcı, Prof, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data are not publicly available due to their containing information that could compromise the privacy of research. However, authors on the subject can be reached.